CLINICAL TRIAL: NCT04708236
Title: A Blinded, Controlled, Escalating Dose Study of ORTD-1 for Treatment of Hospitalized Patients With SARS-CoV-2 (COVID-19) Related Pneumonia.
Brief Title: A Study of ORTD-1 in Patients Hospitalized With COVID-19 Related Pneumonia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: recruitment
Sponsor: Oryn Therapeutics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORTD1-COV-001
Record Dates: First submitted 2021-01-08; First posted 2021-01-13 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: COVID-19 pneumonia; SARS-CoV-2; COVID-19 drug treatment; theta-defensins
MeSH Terms: conditions — COVID-19 | interventions — rhesus-theta-defensin-1

STUDY DESIGN:
Intervention Model Description: Patients will be allocated into 1 of 3 sequential escalating dose cohorts and randomized to ORTD-1 treatment versus vehicle control within each cohort.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ORTD-1 Low dose (Experimental): Arm 1: ORTD-1
  Interventions: Drug: ORTD-1 low dose
- ORTD-1 Mid Dose (Experimental): Arm 2: ORTD-1
  Interventions: Drug: ORTD-1 mid dose
- ORTD-1 High Dose (Experimental): Arm 3 : ORTD-1
  Interventions: Drug: ORTD-1 high dose
- Vehicle Control (Placebo Comparator): Arm 4: Vehicle control
  Interventions: Other: Vehicle control

INTERVENTIONS:
Drug: ORTD-1 low dose — ORTD-1 will be administered intravenously once daily for 5 consecutive days.
  Other Names: Intervention 1
  Arms: ORTD-1 Low dose
Drug: ORTD-1 mid dose — ORTD-1 will be administered intravenously once daily for 5 consecutive days.
  Other Names: Intervention 1
  Arms: ORTD-1 Mid Dose
Drug: ORTD-1 high dose — ORTD-1 will be administered intravenously once daily for 5 consecutive days.
  Other Names: Intervention 1
  Arms: ORTD-1 High Dose
Other: Vehicle control — Vehicle Control will be administered intravenously once daily for 5 consecutive days.
  Other Names: Intervention 2
  Arms: Vehicle Control

SUMMARY:
Evaluate the safety and effect of ORTD-1 on COVID-19 related pneumonia.

DETAILED DESCRIPTION:
This is a randomized, blinded, vehicle-controlled dose-escalation study. Initial enrollment and treatment will be conducted as an inpatient study. Patients will be randomized 2:1, ORTD-1 treatment versus vehicle control. Patients will be allocated into 1 of 3 sequential escalating dose cohorts. Blinded study drug will be infused intravenously once daily for 5 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Positive RT-PCR assay for SARS CoV-2 in a respiratory tract sample
* Hospitalized for COVID-19
* Radiographic diagnosis of pneumonia
* Respiratory insufficiency
* Receiving pharmacologic thromboprophylaxis

Exclusion Criteria:

* Premorbid abnormal pulmonary function or disease
* Concurrent or prior intubation or ventilated support for COVID-19
* Receiving systemic corticosteroids or other immunomodulators or immunosuppressant drugs
* Previous hospitalization for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Through Day 65
  Number of participants with treatment-emergent adverse events
Incidence of laboratory abnormalities | Through Day 65
  Number of participants with Grade 3 or higher laboratory abnormalities
Incidence of anti-drug antibodies | Through Day 65
  Number of participants who develop antibodies to ORTD-1

SECONDARY OUTCOMES:
Proportion of patients requiring intubation | Day 1-65
  The requirement of intubation and invasive ventilation will be assessed for patients at each visit.
Percentage of days requiring supplemental oxygen | Day 1-65
  Percentage of days for which the patient requires supplemental oxygen will be recorded.
Overall survival (OS) | Day 1-65
  Overall survival is defined as the time from enrollment until death from any cause.

OTHER OUTCOMES:
Peripheral blood oxygen levels (SpO2) | Day 1-Day 7, Day 14, Day 21, Day 28, Day 35, Day 65
  SpO2 over time will be measured by pulse oximetry.
IL-6 | Through Day 65
  Level of the inflammatory biomarker IL-6 in blood will be measured.
TNF-alpha | Through Day 65
  Level of the inflammatory biomarker TNF- alpha in blood will be measured.
C-reactive protein | Through Day 65
  Level of the inflammatory biomarker C-reactive protein in blood will be measured.
Serum ferritin | Through Day 65
  Level of serum ferritin in blood will be measured.
D-dimer | Through Day 65
  Level of D-dimer in blood will be measured.
Serum concentration of ORTD-1 (Pharmacokinetics) | Day 1-Day 6, Day 14, Day 21, Day 35, Day 65
  Serum concentration of ORTD-1 will be measured following IV infusion and during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Alpesh Amin, MD, Principal Investigator — Professor & Chair, Department of Medicine University of California, Irvine
Locations (1):
- UC Irvine Medical Center, Orange, California, United States